CLINICAL TRIAL: NCT01946152
Title: A Phase I/II Study of Pomalidomide and Dexamethasone With Growth Factor Support in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Pomalidomide, Dexamethasone, and Filgrastim-sndz in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per PI at time of CR
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0018; NCI-2014-01270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2014-00159; 2013-0018 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Multiple Myeloma-Light Chain Only; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pomalidomide, dexamethasone, filgrastim-sndz) (Experimental): INDUCTION: Patients receive pomalidomide PO daily on days 1-21, dexamethasone PO on days 1, 8, 15, and 22, and filgrastim-sndz SC on days 22-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive lower-dose pomalidomide PO daily on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Biological: Filgrastim-sndz; Other: Laboratory Biomarker Analysis; Drug: Pomalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Biological: Filgrastim-sndz — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Zarxio
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase I/II trial studies the side effects and the best dose of pomalidomide when given together with dexamethasone and filgrastim-sndz and to see how well they work in treating patients with multiple myeloma that has returned or that does not respond to treatment. Pomalidomide may stimulate or suppress the immune system in different ways and may stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Colony-stimulating factors, such as filgrastim-sndz, may increase the production of red and white blood cells and may help the immune system recover from the side effects of pomalidomide and/or dexamethasone. Giving pomalidomide together with dexamethasone and filgrastim-sndz may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of pomalidomide and dexamethasone when given with growth factor support in patients with relapsed and refractory multiple myeloma. (Phase I) II. To evaluate the safety of pomalidomide and dexamethasone at the MTD. (Phase II)

SECONDARY OBJECTIVES:

I. To obtain preliminary estimates of the anti-myeloma activity of higher doses of pomalidomide given with low dose dexamethasone and growth factor support in patients with relapsed and refractory multiple myeloma.

II. Activity will be defined by the overall response rate (ORR); (partial response [PR] or better) and clinical benefit response (CBR) rate (minor response [MR] or better), as well as by the response durability (duration of response [DOR], progression-free survival [PFS], and time to progression [TTP]).

III. To further evaluate the safety of pomalidomide and dexamethasone at the maximum tolerated dose (MTD).

EXPLORATORY OBJECTIVES:

I. To examine the influence of cereblon expression and activation of the wingless-type (Wnt)/beta-catenin pathway on the activity of high dose pomalidomide with low dose dexamethasone.

OUTLINE: This is a phase I, dose-escalation study of pomalidomide followed by a phase II study.

INDUCTION: Patients receive pomalidomide orally (PO) daily on days 1-21, dexamethasone PO on days 1, 8, 15, and 22, and filgrastim-sndz subcutaneously (SC) on days 22-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive lower-dose pomalidomide PO daily on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed and/or refractory multiple myeloma with measurable disease, as defined by one or both of the following (assessed within 14 days prior to initiation of therapy): a) serum myeloma protein (M-protein) >= 0.5 g/d; b) urine Bence-Jones protein >= 200 mg/24 hours
* Patients with light chain only myeloma are eligible; the involved free light chain level >= 100 mg/L with abnormal serum free light chain ratio
* Patients must have prior treatment with >= 2 cycles of lenalidomide and >= 2 cycles of bortezomib (either in separate regimens or as part of the same regimen) (primary refractory of subjects refractory to the most recent regimen are eligible)
* The patient has received =< 5 lines of prior therapy
* Eastern Cooperative Oncology Group performance status 0 - 2
* Serum alanine aminotransferase (ALT) < 3.5 times the upper limit of normal within 7 days of time of consent
* Serum direct bilirubin < 2 mg/dL (34 Omol/L) within 7 days of time of consent
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L within 7 days of time of consent, without granulocyte- colony stimulating factor (G-CSF)
* Hemoglobin > 9 g/dL (80 g/L) within 7 days of time of consent (subjects may be receiving red blood cell transfusions in accordance with institutional guidelines)
* Platelet count > 100 x 10^9/L
* Creatinine clearance > 50 mL/minute within 7 days of time of consent, either measured or calculated using a standard formula (e.g., Cockcroft and Gault)
* Written informed consent in accordance with federal, local, and institutional guidelines
* All study participants must be registered into the mandatory POMALYST (pomalidomide) Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the POMALYST REMS program
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to starting cycle 1 of pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide; FCBP must also agree to ongoing pregnancy testing and follow pregnancy testing requirements as outlined in the POMALYST REMS program; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure

Exclusion Criteria:

* Hypersensitivity to previous lenalidomide or thalidomide
* History of serious allergic reactions to pegfilgrastim or filgrastim
* Chemotherapy (approved or investigational) within 3 weeks prior to signing consent
* Antibody therapy within 6 weeks prior to signing consent
* Radiotherapy to >= 3 sites at the same time within 1 week prior to signing consent
* Immunotherapy within 28 days prior to signing consent
* Pregnant or breast feeding females
* Major surgery within 21 days prior to signing consent
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to signing consent
* Known human immunodeficiency virus infection
* Known active hepatitis B or C infection
* Unstable angina or myocardial infarction within 4 months prior to registration, New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or grade 3 conduction system abnormalities unless subject has a pacemaker
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to signing consent
* Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Significant neuropathy (grades 3 - 4, or grade 2 with pain) within 14 days prior to signing consent
* Subjects with known or likely systemic amyloidosis
* Ongoing graft-vs-host disease
* Any other clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants enrolled, 20 evaluable and 1 screen failure.
Groups:
- Cohort 0: 4 mg of Pomalidomide Daily days 1 - 21. 40 mg Dexamethasone On days 1, 8. 15, 22. 4mcg/kg of Zarxio (G-CSF) Days 22- 28.
- Cohort I; Maximum Tolerated Dose (MTD): 5 mg of Pomalidomide Daily days 1 - 21. 40 mg Dexamethasone On days 1, 8. 15, 22. 4mcg/kg of Zarxio (G-CSF) Days 22- 28.
- Cohort II: 6 mg of Pomalidomide Daily days 1 - 21. 40 mg Dexamethasone On days 1, 8. 15, 22. 4mcg/kg of Zarxio (G-CSF) Days 22- 28.
Period: Overall Study
Arm/Group | Cohort 0 | Cohort I | Cohort II | Maximum Tolerated Dose (MTD)
Started | 3 | 3 | 6 | 8
Completed | 2 | 0 | 0 | 0
Not Completed | 1 | 3 | 6 | 8
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Progression | 0 | 1 | 4 | 7
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Second malignancy | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled on the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 0 | Cohort I | Cohort II | Maximum Tolerated Dose (MTD) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4 | 8
  >=65 years | 2 | 2 | 4 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 3 | 10
  Male | 1 | 0 | 4 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 3 | 0 | 4 | 7 | 14
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 1 | 5
  White | 1 | 3 | 2 | 5 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase I)
Description: Safety and tolerability will be assessed by clinical review of all relevant parameters, including dose limiting toxicities. Toxicity type and severity will be summarized by frequency tables. Maximum tolerated dose defined as the highest dose level in which patients have been treated with less than 2 instances of dose-limiting toxicity (Phase I)
Time Frame: 28 days
Measure: Number; unit: mg
Arm/Group | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 8
mg | 5

2. Primary Outcome: Number of Participants Recommended Phase II Dose of Pomalidomide and Dexamethasone, When Both Agents Are Administered Together With Granulocyte-colony Stimulating Factor (Filgrastim) (Phase I)
Time Frame: Up to 28 days
Population: Data provided for the Participants who received MTD
Measure: Count of Participants; unit: Participants
Arm/Group | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 8
Participants | 8

3. Secondary Outcome: Number of Participants With Best Overall Response Defined Using the International Myeloma Working Group Uniform Response Criteria (IMWG-URC)
Description: Per International Myeloma Working Group Uniform Response Criteria (IMWG-URC): Complete Response (CR), Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow; Very Good Partial Response (VGPR): Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% reduction in serum M-protein with urine M-protein <100 mg/24 hours; Partial Response (PR), > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h; Stable Disease (SD) = CR + PR.
Time Frame: After 112 days (4 courses) of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 | Cohort I | Cohort II | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 3 | 3 | 6 | 8
Participants
  Partial Response | 1 | 2 | 3 | 6
  Progression Disease | 0 | 1 | 1 | 0
  Stable Disease | 1 | 0 | 1 | 1
  Complete Response | 0 | 0 | 0 | 0
  Very Good Partial Response (VGPR) | 1 | 0 | 0 | 1
  Non evaluable | 0 | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Progression-free Survival
Time Frame: Up to 6 years
Population: Data provided for the Participants who received MTD
Measure: Count of Participants; unit: Participants
Groups:
- Maximum Tolerated Dosage (MTD): 5 mg of Pomalidomide Daily days 1 - 21. 40 mg Dexamethasone On days 1, 8. 15, 22. 4mcg/kg of Zarxio (G-CSF) Days 22- 28.
Arm/Group | Maximum Tolerated Dosage (MTD)
Number analyzed (Participants) | 8
Participants | 3

ADVERSE EVENTS:
Time Frame: From start of treatment until 30 days after last dose, up to 6 years
Groups:
- Cohort 1; Maximum Tolerated Dose (MTD): 5 mg of Pomalidomide Daily days 1 - 21. 40 mg Dexamethasone On days 1, 8. 15, 22. 4mcg/kg of Zarxio (G-CSF) Days 22- 28.
- Cohort 2: 6 mg of Pomalidomide Daily days 1 - 21. 40 mg Dexamethasone On days 1, 8. 15, 22. 4mcg/kg of Zarxio (G-CSF) Days 22- 28.
Arm/Group | Cohort 0 | Cohort 1 | Cohort 2 | Maximum Tolerated Dose (MTD)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 2/6 | 1/8
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/6 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0 (N=3) | Cohort 1 (N=3) | Cohort 2 (N=6) | Maximum Tolerated Dose (MTD) (N=8)
Sinusitis (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Febrile Neutropenia (Infections and infestations) | 0 | 0 | 1 | 0
Squamous Cell CA (General disorders) | 0 | 0 | 1 | 0
Fall/Hip Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Fecal Incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Syncope (Cardiac disorders) | 0 | 0 | 0 | 1
Dyspnea (Cardiac disorders) | 0 | 0 | 0 | 1
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0 (N=3) | Cohort 1 (N=3) | Cohort 2 (N=6) | Maximum Tolerated Dose (MTD) (N=8)
Febrile Neutropenia (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0
Secondary Cancers (General disorders) | 0 | 0 | 0 | 2
Pain Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2 | 0
Chest Pain (Cardiac disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Myalgia (General disorders) | 0 | 1 | 0 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Anemia (Immune system disorders) | 0 | 1 | 0 | 0
Skin Disorders (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT01946152/Prot_SAP_000.pdf